CLINICAL TRIAL: NCT02921867
Title: A Randomized Trial on the Effect of Simulation-based Diagnostic Abdominal Ultrasound Training
Brief Title: A Trial on the Effect of Simulation-based Diagnostic Abdominal Ultrasound Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mia Louise Østergaard, MD, PhD researchfellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Abd.Sim.Training.RT
Record Dates: First submitted 2016-09-21; First posted 2016-10-03 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Pathology
Keywords: ultrasound; radiology; simulation; abdominal ultrasound; medical education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Simulation-based training in nine modules with optional training times and ending with an obligatory certification test before traditional training is started. Traditional training time unaltered: six weeks.
  Interventions: Other: Simulation-based training
- Traditional training (No Intervention): Six weeks focused stay at an ultrasound ward with day to day one-on-one supervision (current practise)

INTERVENTIONS:
Other: Simulation-based training — The simulation-based training will consist of nine modules that can be trained in random order and training periods within the eight weeks before clinical training starts.
  Arms: Intervention group

SUMMARY:
The investigators hypothesise that simulation-based training will have initial educational benefits and in coherence with the traditional apprenticeship model will heighten the educational end-level: That training on the simulator before clinical education will prepare the trainee for practice and thereby support more effective learning.

DETAILED DESCRIPTION:
This study will be registered at ClincalTrials.gov and reported according to the CONSORT statement.

Setting: Clinical training will forego unaltered as current practice at the department of the individual resident's employment. The simulated training will be held as individual training sessions on the Schallware Ultrasound simulator (station 64; version 010013) placed at the Copenhagen Academy for Education and Simulation (CAMES), Rigshospitalet. Testing will be done on both the simulator at the Simulationcentre at Rigshospitalet, CAMES and on real life patients in the departments of radiology where the residents are employed.

Population: Participants are residents embarking on the first year of their specialized radiological training before any formalized ultrasound training. Enrollment is voluntary and in collaboration with their department of employment.

Intervention and controlled conditions:

A total of 22 residents at the beginning of their specialized radiological education and before their focused ultrasound training are randomised for two educational groups.

The simulation-based training modules will be in a recommend but not mandatory order starting with a general organ-identifying module and continuing with range of pathology modules with headlines: Introduction, Liver I, Liver II, Biliary System, Pancreas and Spleen, Urinary System, Vessels, Other Findings, and Mixed Cases.

The clinical part of training will forego unaltered for both groups for six weeks and all participants will fill out a log of all scans performed and when supervised the supervisor will score their scans using the OSAUS score.

The reviewer scoring the simulation-based test will be blinded. It is not possible to blind the reviewers of the clinical score (OSAUS) as it is the residents' clinical supervisors.

ELIGIBILITY:
Inclusion Criteria:

* Fluent oral and written Danish or English.

Exclusion Criteria:

* Clinical ultrasound training or completed ultrasound courses with or without simulation training for more than one week in total prior to enrollment.
* Failure to complete simulation-based training or pass the simulation-based diagnostic ultrasound test. Failure to complete the logbook.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
All participants in both groups will be scored during their clinical ultrasound training by their supervising physicians using Objective Structured Assessment of Ultrasound Skills (OSAUS) | Enrollment will forego until 22 residents in total has been enrolled; expectantly in 9-12 month..

CONTACTS AND LOCATIONS:
Overall Officials: Mia L Østergaard, MD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Copenhagen University hospital, Rigshospitalet, Copenhagen, Copenhagen O, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Todsen T, Tolsgaard MG, Olsen BH, Henriksen BM, Hillingso JG, Konge L, Jensen ML, Ringsted C. Reliable and valid assessment of point-of-care ultrasonography. Ann Surg. 2015 Feb;261(2):309-15. doi: 10.1097/SLA.0000000000000552. PMID 24509198
- [Derived] Ostergaard ML, Rue Nielsen K, Albrecht-Beste E, Kjaer Ersboll A, Konge L, Bachmann Nielsen M. Simulator training improves ultrasound scanning performance on patients: a randomized controlled trial. Eur Radiol. 2019 Jun;29(6):3210-3218. doi: 10.1007/s00330-018-5923-z. Epub 2019 Jan 7. PMID 30617476